CLINICAL TRIAL: NCT01593969
Title: A Randomised Controlled Trial of n-3 Polyunsaturated Fatty Acid-Enriched Therapeutic Food for Childhood Severe Malnutrition
Brief Title: A Trial of n-3 PUFA-Enriched Ready to Use Therapeutic Food for Childhood Severe Malnutrition
Acronym: Njugu Plus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSC 2157; OPP1046183 (Other Grant/Funding Number: The Bill & Melinda Gates Foundation)
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Severe Acute Malnutrition
Keywords: Essential Fatty Acid; Seed oil; Fish oil; Dietary deficiency
MeSH Terms: conditions — Severe Acute Malnutrition; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard RUTF (Active Comparator): Standard RUTF given according to National Guidelines
  Interventions: Dietary Supplement: Standard RUTF
- RUTF/Flax Oil (Experimental): RUTF/Flax Oil is reformulated RUTF to increase n3 content
  Interventions: Dietary Supplement: RUTF/Flax Oil
- RUTF/Flax Oil plus additional Fish Oil (Experimental): RUTF/Flax Oil plus additional Fish Oil is RUTF reformulated to increase n3. Fish oil to provide long chain n3
  Interventions: Dietary Supplement: RUTF/Flax Oil plus additional Fish Oil

INTERVENTIONS:
Dietary Supplement: RUTF/Flax Oil — Ready to Use Therapeutic Food
  Arms: RUTF/Flax Oil
Dietary Supplement: RUTF/Flax Oil plus additional Fish Oil — Ready to Use Therapeutic Food
  Arms: RUTF/Flax Oil plus additional Fish Oil
Dietary Supplement: Standard RUTF — Standard formulation RUTF given according to National Guidelines
  Arms: Standard RUTF

SUMMARY:
The investigators will perform a randomised controlled trial of the provision of food designed for rehabilitation of malnourished children that is supplemented with n-3 fatty acids compared to usual composition. The investigators want to see whether the provision of such a food normalises the deficiencies in essential fatty acids observed in severely malnourished children faster than standard composition.

DETAILED DESCRIPTION:
Randomized controlled trial of n-3 Polyunsaturated Fatty Acid-Enriched Therapeutic Food for Severe Malnutrition.

Description of Study Design: Randomized Controlled Trial

Study Duration: 6 months (Trial); 12 months (All trial-related activities)

Description of Intervention: Provision of ready to use food (RUTF) enriched with flax seed oil, with or without fish oil, compared to conventional-composition RUTF. Interventional product will be given until nutritional recovery to a maximum of 12 weeks.

Design: Flax-enriched or standard RUTF allocation is randomised and double blind. Fish oil allocation is randomised within those receiving flax-enriched RUTF and is open label.

Location: Kilifi District, coastal Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 5 years old
* Provision of informed consent
* Severe malnutrition (one or more of mid-upper arm circumference <11.5cm, weight for height z score <-3, or nutritional oedema)
* Stabilised and eligible to receive RUTF according to national guidelines

Exclusion Criteria:

* Known HIV disease, tuberculosis or other chronic infection*
* Known allergy or hypersensitivity to any of the product ingredients

  * Chronic infections such as HIV and tuberculosis and their treatments are likely to cause alterations in lipid metabolism that may confound interpretation of this pilot trial. national guidelines recommend offering provider-initiated testing for HIV for all severely malnourished children, and referral for comprehensive care in the case of a positive test.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Total long chain PUFA in erythrocyte membranes at 3 months | 3 months
  Total long chain PUFA in erythrocyte membranes at 3 months

SECONDARY OUTCOMES:
Ratio of n-6:n-3 PUFA in erythrocyte membranes at 3 months | 3 months
  Ratio of n-6:n-3 PUFA in erythrocyte membranes at 3 months
Total long chain PUFA in CD3 cell membranes at 3 months | 3 months
  Total long chain PUFA in CD3 cell membranes at 3 months
Ratio of n-6:n-3 PUFA in CD3 cell membranes at 3 months | 3 months
  Ratio of n-6:n-3 PUFA in CD3 cell membranes at 3 months
Total long chain PUFA in plasma at 3 months | 3 months
  Total long chain PUFA in plasma at 3 months
Ratio of n-6:n-3 PUFA in plasma at 3 months | 3 months
  Ratio of n-6:n-3 PUFA in plasma at 3 months
Change in weight for height z score between baseline and 3 months | 3 months
  Change in weight for height z score between baseline and 3 months
Change in mid upper arm circumference between baseline and 3 months | 3 months
  Change in mid upper arm circumference between baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James A Berkley, FRCPCH, Principal Investigator — KEMRI-Wellcome Trust Collaborative Research Program
Locations (1):
- Kilifi District Hospital, Kilifi, Coast, Kenya

REFERENCES:
- [Derived] Jones KD, Ali R, Khasira MA, Odera D, West AL, Koster G, Akomo P, Talbert AW, Goss VM, Ngari M, Thitiri J, Ndoro S, Knight MA, Omollo K, Ndungu A, Mulongo MM, Bahwere P, Fegan G, Warner JO, Postle AD, Collins S, Calder PC, Berkley JA. Ready-to-use therapeutic food with elevated n-3 polyunsaturated fatty acid content, with or without fish oil, to treat severe acute malnutrition: a randomized controlled trial. BMC Med. 2015 Apr 23;13:93. doi: 10.1186/s12916-015-0315-6. PMID 25902844